CLINICAL TRIAL: NCT04340219
Title: A Prospective Cohort Study Investigating Oncology-patient-reported Anxiety, Mood, and Quality of Life During the COVID-19 Pandemic (ONCOVID Trial)
Brief Title: Oncology-patient-reported Anxiety, Mood, and QoL During the COVID-19 Pandemic
Acronym: ONCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07505-LGE
Record Dates: First submitted 2020-03-31; First posted 2020-04-09 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: COVID-19; Quality of Life; Anxiety; Stress; Mood; DASS-21; WHOQOL-BREF; CPDI
MeSH Terms: conditions — Neoplasms; COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients: Participants complete a survey consisting of sociodemographic information and self-administered questionnaires (CPDI, DASS-21, and WHOQOL-BREF).
  Interventions: Other: Survey administration

INTERVENTIONS:
Other: Survey administration — Covid-19 Peritraumatic Distress Index, Depression Anxiety Stress Scale-21, WHO Quality of Life-BREF

SUMMARY:
ONCOVID is a prospective cohort study investigating oncology-patient-reported anxiety, mood, and quality of life during the COVID-19 pandemic. Participants complete a survey consisting of sociodemographic information and self-administered questionnaires (COVID-19 Peritraumatic Distress Index, Depression Anxiety Stress Scale-21, and WHO Quality of Life-BREF). Data collection occurs at baseline and follow-up surveys are performed after 6, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically confirmed cancer
* Receive systemic therapy (including chemotherapy, targeted small-molecule therapy, anticancer monoclonal antibody, immunotherapy, endocrine therapy, or investigational agent) (either exclusively or in combination with other anticancer therapy) between February 14, 2020 and March 31, 2020 (Note: Patients whose systemic treatment administration was initially planned for this period but was modified, delayed, stopped, or withheld due to COVID-19 measures are also eligible for inclusion)

Exclusion Criteria:

* Insufficient understanding of the Dutch language
* Severe cognitive impairment
* Acute psychiatric crisis
* Not able to give informed consent
* Confirmed or clinically suspected COVID-19
* Endocrine therapy in (neo)adjuvant setting (Note: Patients whose (neo)adjuvant systemic treatment was initially planned as chemotherapy, targeted small-molecule therapy, anticancer monoclonal antibody, immunotherapy, or investigational agent (either exclusively or in combination in combination with other anticancer therapy) but was modified to endocrine therapy due to COVID-19 measures are also eligible for inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing systemic treatment at the Medical Oncology Department between February 14 and March 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Distress at baseline measured by the COVID-19 Peritraumatic Distress Index (CPDI); in terms of proportions (0-28 vs ≥ 29). | Week 0
Depression at baseline measured by the 7-item depression subscale of the 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression); in terms of proportions (0-4 vs ≥ 5). | Week 0
Anxiety at baseline measured by the 7-item anxiety subscale of the DASS-21 (DASS-21-Anxiety); in terms of proportions (0-3 vs ≥ 4). | Week 0
Stress at baseline measured by the 7-item stress subscale of the DASS-21 (DASS-21-Stress); in terms of proportions (0-7 vs ≥ 8). | Week 0

SECONDARY OUTCOMES:
Distress measured at baseline by the CPDI; in terms of continuous values. | Week 0
Depression at baseline measured by the DASS-21-Depression; in terms of continuous values. | Week 0
Anxiety at baseline measured by the DASS-21-Anxiety; in terms of continuous values. | Week 0
Stress at baseline measured by the DASS-21-Stress; in terms of continuous values. | Week 0
Domain-specific quality of life at baseline measured by the 7-item physical health domain of the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire (WHOQOL-BREF-Physical health); in terms of continuous values. | Week 0
Domain-specific quality of life at baseline measured by the 6-item psychological health domain of the WHOQOL-BREF questionnaire (WHOQOL-BREF-Psychological health); in terms of continuous values. | Week 0
Domain-specific quality of life at baseline measured by the 3-item social relationships domain of the WHOQOL-BREF questionnaire (WHOQOL-BREF-Social relationships); in terms of continuous values. | Week 0
Domain-specific quality of life at baseline measured by the 8-item environment domain of the WHOQOL-BREF questionnaire (WHOQOL-BREF-Environment); in terms of continuous values. | Week 0
Overall perception of quality of life and overall perception of health at baseline measured by the two items from the Overall QOL and General Health in the WHOQOL-BREF questionnaire-in terms of continuous values. | Week 0
Change from baseline in distress measured by CDPI; in terms of continuous values. | 24 weeks
Change from baseline in depression measured by the DASS-21-Depression; in terms of continuous values. | 24 weeks
Change from baseline in anxiety measured by the DASS-21-Anxiety; in terms of continues values. | 24 weeks
Change from baseline in stress measured by the DASS-21-Stress; in terms of continuous values. | 24 weeks
Change from baseline in domain-specific quality of life at baseline measured by the WHOQOL-BREF-Physical health; in terms of continuous values. | 24 weeks
Change from baseline in domain-specific quality of life at baseline measured by the WHOQOL-BREF-Psychological health; in terms of continuous values. | 24 weeks
Change from baseline in domain-specific quality of life measured by the WHOQOL-BREF-Social relationship; in terms of continuous values. | 24 weeks
Change from baseline in domain-specific quality of life measured by the WHOQOL-BREF-Environment; in terms of continuous values. | 24 weeks
Change from baseline in overall perception of quality of life and overall perception of health measured by the 2 items from the Overall QOL and General Health in the WHOQOL-BREF questionnaire; in terms of continuous values. | 24 weeks
The real-life impact of COVID-19 on systemic treatment administration will be assessed using descriptive statistics | Week 0-6-12-24

CONTACTS AND LOCATIONS:
Overall Officials: Hannelore Denys, MD, PhD, Principal Investigator — Medical Oncologist
Locations (1):
- University Hospital Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No